CLINICAL TRIAL: NCT05225519
Title: Effects of Far Infrared Radiation on Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Academic Center (2CA-Braga) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FibroFIR
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Usage of a long-sleeved white shirt impregnated with a long-infrared irradiating bioceramic for a period of 12 weeks.
  Interventions: Device: long-sleeved white shirt impregnated with a long-infrared irradiation
- Placebo arm (Placebo Comparator): Usage of a long-sleeve white shirt (similar to the one in the experimental arm) but with no long-infrared technology for a period of 12 weeks.
  Interventions: Device: long-sleeved white shirt

INTERVENTIONS:
Device: long-sleeved white shirt impregnated with a long-infrared irradiation — Usage of an experimental shirt for a period of 12 weeks.
  Arms: Experimental arm
Device: long-sleeved white shirt — Usage of an experimental shirt for a period of 12 weeks.
  Arms: Placebo arm

SUMMARY:
This study aimed to evaluate the effectiveness of infrared radiation in improving the various symptoms of fibromyalgia syndrome, by using a long-sleeved white shirt impregnated with a long-infrared irradiating bioceramic, as well as the adherence to it and its applicability in daily routines.

A prospective, experimental, randomized, and double-blind study was carried. The study was implemented over 7 months, with a total of 5 visits for each patient. Participants were randomly allocated in experimental or control group. Those included in the experimental group received a shirt impregnated with ceramic emitting long infrared waves while participants in the placebo group received an exactly looking shirt, but not impregnated with ceramic emitting long infrared waves. Each visit comprised clinical evaluation and self-report scales filling (WPS, SS and FIQR scales).

ELIGIBILITY:
Inclusion Criteria:

* age superior to 18 years-old
* ability to freely sign the informed consent form
* generalized pain index scores (WPI ≥ 7 and SS score ≥ 5, or WPI ≥ 3 and ≤ 6 with SS ≥ 9, presence of abdominal pain and / or with depression and / or headache, in the last 6 months, at the screening consultation).

Exclusion Criteria:

* dermatological diseases
* Other rheumatic and /or autoimmune diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
WPI | Change between baseline and after 4, 8 and 12 weeks of wearing the shirt.
  The widespread pain index (WPI) is a 19-point checklist (score range: 0-19) that assesses the presence of pain or tenderness score means (within the prior seven days) in 19 specific areas of the body; each affected area receives one point.
SS | Change between baseline and after 4, 8 and 12 weeks of wearing the shirt.
  The symptom severity score (SS) quantifies symptom severity on a 0-12 scale by assessing problems with fatigue, cognitive dysfunction and unrefreshed sleep over the past week. These scores are summed for a measure of the physician's impression of the number of somatic symptoms the patient has on a 0-3 scale.

SECONDARY OUTCOMES:
FIQR | Change between baseline and after 4, 8 and 12 weeks of wearing the shirt.
  Revised Fibromyalgia Impact Questionnaire (FIQR) is a 21-item self-administered questionnaire. All items are visual analogue scales with 11 boxes discreetly scoring from 0 to 10 with 10 being 'worst'. All questions are framed in the context of the past 7 days.
Tender Points | Change between baseline and after 4, 8 and 12 weeks of wearing the shirt.
  Number of tender points at the moment.
EQ-5D | Change between baseline and after 4, 8 and 12 weeks of wearing the shirt.
  EQ-5D is a standardized measure of health-related quality of life. EQ-5D assesses health status in terms of five dimensions of health (mobility, self-care, usual activities, pain and discomfort, and anxiety and depression).

CONTACTS AND LOCATIONS:
Locations (1):
- 2CA-Braga, Braga, Portugal

IPD SHARING:
Plan to Share IPD: No